CLINICAL TRIAL: NCT02167451
Title: Maraviroc as Graft Versus Host Disease Prophylaxis in Pediatric and Adult Stem Cell Transplant Recipients
Brief Title: Maraviroc as GVHD Prophylaxis in Transplant Recipients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow recruitment and no further drug supply
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-1221
Record Dates: First submitted 2014-06-13; First posted 2014-06-19 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Diagnoses That Require Stem Cell Transplant; Graft Versus Host Disease (GVHD)
Keywords: stem cell transplant; GVHD prevention
MeSH Terms: conditions — Graft vs Host Disease | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maraviroc (Experimental): Maraviroc administration will start on day -3 and will end on day +30 after stell cell transplant, making the total number of days of drug administration 34 days. Maraviroc will be administered twice daily orally or via enteral tube. Dosing of Maraviroc will be based on body surface area (starting with 100mg twice a day for BSA of 0.2 and up to 300mg twice a day for BSA greater than 1.73).
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc
  Other Names: Selzentry

SUMMARY:
The purpose is to determine if the addition of Maraviroc to a standard transplant regimen will reduce the incidence of graft versus host disease in children and young adults after a stem cell transplant.

DETAILED DESCRIPTION:
In the first stage, drug levels will be obtained to establish appropriate dosing. In the second stage of the study the investigators will study the effects of using Maraviroc in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5 years and </= 40 years
* All diagnoses
* Peripheral blood stem cells, marrow or cord blood
* All conditioning regimens
* Patient must be planned to receive a calcineurin inhibitor (cyclosporine or tacrolimus) together with steroid, methotrexate or mycophenolate mofetil as GVHD prophylaxis.

Exclusion Criteria:

* Documented anaphylaxis to Maraviroc
* Ex vivo T-cell (type of white blood cell) depleted grafts
* Abnormal Alanine Aminotransferase (ALT) (>/=10X ULN) on day -3. (Assessed at study enrollment and confirmed again prior to the first dose of maraviroc.)

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Khandelwal, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc: Maraviroc administration will start on day -3 and will end on day +30 after stell cell transplant, making the total number of days of drug administration 34 days. Maraviroc will be administered twice daily orally or via enteral tube. Dosing of Maraviroc will be based on body surface area (starting with 100mg twice a day for BSA of 0.2 and up to 300mg twice a day for BSA greater than 1.73).
  Maraviroc
Period: Overall Study
Arm/Group | Maraviroc
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: not different
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Maraviroc
Description: The ability to administer twice daily oral maraviroc in children and adults undergoing stem cell transplant in addition to routine standard graft versus host disease prophylaxis.
Time Frame: Up to day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
Participants | 23

2. Primary Outcome: GVHD Incidence
Description: Incidence of GVHD by day+100
Time Frame: By day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
Participants | 11

3. Primary Outcome: Area Under The Concentration-Time Curve (AUC) of Maraviroc
Description: pK target >100ng/ml at day zero at the following time points : before the dose and 1, 2, 4, 6, 8, and 12 hours after maraviroc administration
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: hour *ng/mL
Arm/Group | Maraviroc
Number analyzed (Participants) | 12
hour *ng/mL | 4805 (3265)

4. Primary Outcome: Incidence of Visceral GVHD
Description: determine the number of patients who develop visceral GVHD by day+100
Time Frame: day+100
Population: all patients enrolled on trial
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
Participants | 6

5. Primary Outcome: Area Under The Concentration-Time Curve (AUC) of Maraviroc
Description: pK target >100ng/ml at day 10 at the following time points : before the dose and 1, 2, 4, 6, 8, and 12 hours after maraviroc administration
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Maraviroc
Number analyzed (Participants) | 12
hour*ng/mL | 5917 (4048)

6. Secondary Outcome: Overall Survival
Description: Overall survival for patients who were enrolled and received maraviroc
Time Frame: By day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
Participants | 27

7. Secondary Outcome: Graft Failure
Description: Failure to engraft and loss of graft.
Time Frame: By day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
Participants | 4

8. Secondary Outcome: Primary Disease Relapse
Time Frame: By day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
Participants | 0

9. Secondary Outcome: Toxicities
Description: Incidence of toxicities due to drug
Time Frame: Up to day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
Participants | 0

10. Secondary Outcome: Infectious Complications
Description: Infections complications which include asymptomatic viremias for EBV, Adenovirus, CMV, and/or viral disease, bacterial and fungal infections as documented by blood cultures.
Time Frame: Up to day +100
Measure: Number; unit: patients
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
patients
  bacterial infections | 11
  Fungal infections | 2
  CMV | 5
  EBV | 4
  Adenovirus | 2
  Bk viremia | 5

11. Secondary Outcome: Time to Neutrophil
Description: Neutrophil engraftment is defined as the first of three consecutive measurements of ANC>500mcL over 3 or more days.
Time Frame: Up to day +100
Measure: Median (Full Range); unit: days
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
days | 11 [8 to 16]

12. Secondary Outcome: Time to Platelet Engraftment
Description: Time to achieve platelets count of 20,000 without transfusions
Time Frame: days
Measure: Median (Full Range); unit: days
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
days | 18 [15 to 38]

ADVERSE EVENTS:
Time Frame: day+ 100 after BMT or 30 days after last maraviroc administration if patients withdrew from study
Arm/Group | Maraviroc
All-Cause Mortality (participants affected / at risk) | 4/31
Serious Adverse Events (participants affected / at risk) | 11/31
Other Adverse Events (participants affected / at risk) | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc (N=31)
TMA (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1)
Sinusoidal Obstructive Syndrome (Investigations) | 3 (3)
Infection- Disseminated Adenoviremia (Infections and infestations) | 2 (2)
Infection- Enterobacter Aerogenes Baceteremia (Infections and infestations) | 1 (1)
Infection-Enterococcus Bacteremia (Infections and infestations) | 3 (3)
Infection-Citrobacter and Klebsiella Bacteremia (Infections and infestations) | 1 (1)
Infection- Klebsiella Pneumonia Bacteremia (Infections and infestations) | 1 (1)
Infection- Staphylococcus Aureus Bacteremia (Infections and infestations) | 3 (3)
Infection- CMV Viremia (Infections and infestations) | 1 (1)
Immune System Other (Engraftment Syndrome) (Immune system disorders) | 2 (2)
Allergic Reaction (Angioedema) (Immune system disorders) | 1 (1) — Angioedema was not due to maraviroc as drug was stopped . This was experienced post anesthesia .
Blood Bilirubin- Increased (Investigations) | 5 (6)
Altered mental status (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis due to CMV (Respiratory, thoracic and mediastinal disorders) | 1 (1)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc (N=31)
anemia (Blood and lymphatic system disorders) | 6 (8)
TMA/HUS (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 6 (6)
Fever (General disorders) | 1 (1)
Sinusoidal Obstructive Syndrome (Hepatobiliary disorders) | 1 (1)
Allergic reaction to Ambisome (Immune system disorders) | 1 (1)
Anaphylaxis to Cyclosporine (Immune system disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
CMV viremia (Infections and infestations) | 1 (1)
catheter related infection ( MSSA bacteremia, staph aureus and bacillus) (Infections and infestations) | 1 (1)
Adenovirus in stool (Infections and infestations) | 1 (1)
Adenovirus in blood (Infections and infestations) | 2 (2)
BK viremia (Infections and infestations) | 1 (1)
Moraxella nonliquefaciens infection in blood (Infections and infestations) | 1 (1)
HHV6 blood (Infections and infestations) | 1 (1)
Streptococcus infection in blood (Infections and infestations) | 1 (1)
Klebsiella oxytoca infection in blood (Infections and infestations) | 1 (1)
Candida in blood (Infections and infestations) | 1 (1)
Escherichia Coli in blood (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 12 (12)
hemoglobin decreased (Investigations) | 1 (1)
WBC decreased (Investigations) | 9 (9)
Platelet count decreased (Investigations) | 10 (12)
Lymphocyte count decreased (Investigations) | 5 (13)
ALT increased (Investigations) | 2 (2)
AST increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 4 (4)
creatinine increased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02167451/Prot_SAP_000.pdf